CLINICAL TRIAL: NCT05243680
Title: A Multi-centre, Single Arm, Open-label Extension Study to Evaluate the Long-term Safety of GSK3511294 (Depemokimab) in Adult and Adolescent Participants With Severe Asthma With an Eosinophilic Phenotype From Studies 206713 or 213744
Brief Title: An Open-Label Extension Study of GSK3511294 (Depemokimab) in Participants Who Were Previously Enrolled in 206713 (NCT04719832) or 213744 (NCT04718103)
Acronym: AGILE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212895; 2023-505203-23-01 (Other: EU-CT)
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: GSK3511294; Depemokimab; Asthma; Long-term safety; Open-label
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants diagnosed with asthma receiving GSK3511294 (Depemokimab) (Experimental)
  Interventions: Biological: GSK3511294 (Depemokimab)

INTERVENTIONS:
Biological: GSK3511294 (Depemokimab) — GSK3511294 (Depemokimab) will be administered using a pre-filled safety syringe.

SUMMARY:
The purpose of this open-label 12-month extension study is to continue to characterize the long-term safety, efficacy and immunogenic profile of GSK3511294 (Depemokimab) in participants with severe asthma with an eosinophilic phenotype following completion of clinical studies 206713 or 213744.

ELIGIBILITY:
Inclusion criteria:

* Participants who completed the double-blind study intervention treatment during Study 206713 or Study 213744.
* Participants capable of giving signed informed consent/assent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. In France, a participant will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion criteria:

* Clinically significant change in health status during Study 206713 or Study 213744 which in the opinion of the investigator would make the participant unsuitable for participation in this study.
* A current malignancy or a malignancy that developed during Study 206713 or Study 213744 (participants who had localized carcinoma of the skin that was resected for cure will not be excluded).
* Participants who have other clinically significant medical conditions uncontrolled with Standard of Care (SoC) therapy not associated with Asthma, for example (e.g.), uncontrolled cardiovascular disease or ongoing active infectious disease which in the opinion of the investigator makes them unsuitable for the study.
* Participants with known parasitic (helminth) infections within 6 months prior to Visit 1 will be excluded from the study or required to be adequately treated for helminth infections before initiation of GSK3511294.
* Participants who meet the following based on results of Week 48 assessment from Study 206713 or Study 213744 or from a later result:

  1. Alanine aminotransferase (ALT) greater than (>)2 times upper limit of normal (ULN).
  2. Total bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin less than [<] 35 percent [%]).
  3. Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice.
* Participants with current diagnosis of vasculitis. Participants with high clinical suspicion of vasculitis at screening will be evaluated and current vasculitis must be excluded prior to enrolment.
* Electrocardiogram (ECG) assessment: QTc corrected by Fridericia's formula (QTcF) greater than or equal to (>=)450 milliseconds (msec) or QTcF >=480 msec for participants with Bundle Branch Block at Visit 1.
* Current smokers.
* Participants with allergy/intolerance to the excipients of GSK3511294, a monoclonal antibody, or biologic.
* Participants who are pregnant or breastfeeding. Participants should not be enrolled if they plan to become pregnant during the time of study participation.
* Participants who for any reason permanently discontinued study treatment in the previous study 206713/213744 will be excluded from this study.
* Other investigational product/clinical study:

  1. Participants who have received treatment with an investigational agent (biologic or non-biologic) within the past 30 days or 5 drug half-lives whichever is longer, prior to the first dose, other than Study 206713/213744 study treatment. The term "investigational" applies to any drug not approved for sale for the disease/indication to treat in the country in which it is being used or investigational formulations of marketed products.
  2. Participants who are currently participating in any other interventional clinical study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (116):
- United States (26):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Lancaster, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Lafayette, Colorado
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Loxahatchee Groves, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Northfield, New Jersey
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, DuBois, Pennsylvania
  - GSK Investigational Site, Allen, Texas
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Bellingham, Washington
- Australia (2):
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, South Brisbane, Queensland
- Canada (4):
  - GSK Investigational Site, Sherwood Park, Alberta
  - GSK Investigational Site, Kamloops, British Columbia
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Ottawa, Ontario
- China (15):
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Haikou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Hefei
  - GSK Investigational Site, Hohhot
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Shenyang
  - GSK Investigational Site, Ürümqi
  - GSK Investigational Site, Wenzhou
  - GSK Investigational Site, Wuhan
  - GSK Investigational Site, Xuzhou
- Czechia (6):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Strakonice
  - GSK Investigational Site, Tábor
  - GSK Investigational Site, Teplice
- France (4):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Cholet
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Strasbourg
- Germany (7):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Koblenz
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Magdeburg
  - GSK Investigational Site, Neu-Isenburg
- Hungary (3):
  - GSK Investigational Site, Gödöllő
  - GSK Investigational Site, Mosonmagyaróvár
  - GSK Investigational Site, Szigetvár
- Italy (11):
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Foggia
  - GSK Investigational Site, Messina
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Monserrato CA
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Rozzano MI
  - GSK Investigational Site, Siena
  - GSK Investigational Site, Varese
- Japan (13):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Tokyo
- Poland (8):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Strzelce Opolskie
- Spain (10):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Benalmádena
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- Taiwan (2):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
- United Kingdom (5):
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Chertsey
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who successfully completed treatment in studies 206713 (NCT04719832), and 213744 (NCT04718103) were eligible to continue their treatment in this open-label extension study 212895.
Pre-assignment Details: A total of 641 participants were enrolled in this study, however only 629 participants were included in Safety Analysis Set (SAS) (as 12 participants were excluded from the SAS due to data integrity and good clinical practices [GCP] violations). SAS included all participants who received at least one dose of open-label GSK3511294 in this extension study, excluding the participants from the sites with data integrity and GCP violation issues.
Groups:
- Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study: Participants who had previously received placebo in the 206713 (NCT04719832) and 213744 (NCT04718103) were enrolled in this extension study. Participants received a 100 milligram (mg) dose of GSK3511294 as a subcutaneous (SC) injection once on Week 0 (visit 1) and on Week 26 (visit 6) in this extension study. Participants were to be maintained on their existing Baseline maintenance asthma standard of care (SOC) treatment throughout the study.
- GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study: Participants who had previously received GSK3511294 100 mg subcutaneously (SC) in the 206713 (NCT04719832) and 213744 (NCT04718103) were enrolled in this extension study. Participants received a 100 mg dose of GSK3511294 as a SC injection once on Week 0 (visit 1) and on Week 26 (visit 6) in this extension study. Participants were to be maintained on their existing Baseline maintenance asthma SOC treatment throughout the study.
Period: Overall Study
Arm/Group | Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study | GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study
Started (Enrolled) | 214 | 427
Safety Analysis Set | 210 | 419
Completed | 199 | 403
Not Completed | 15 | 24
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 5 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 3 | 10
Not completed — Data integrity and GCP violations | 4 | 8

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for the Safety Analysis Set which included all participants who received at least one dose of open-label GSK3511294 in this extension study, excluding the participants from the sites with data integrity and GCP violation issues.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study | GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study | Total
Number analyzed (Participants) | 210 | 419 | 629
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (15.84) | 55.5 (14.84) | 54.8 (15.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 248 | 376
  Male | 82 | 171 | 253
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 169 | 321 | 490
  ASIAN | 35 | 81 | 116
  AMERICAN INDIAN OR ALASKA NATIVE | 1 | 2 | 3
  BLACK OR AFRICAN AMERICAN | 5 | 15 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: Up to Week 56
Population: Safety Analysis Set included all participants who received at least one dose of open-label GSK3511294 excluding the participants from the sites with data integrity and GCP violation issues.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study | GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study
Number analyzed (Participants) | 210 | 419
Participants
  Any AEs | 147 | 301
  Any SAEs | 21 | 38

2. Primary Outcome: Number of Participants With Worst Case Post-Baseline Positive Anti-GSK3511294 Antibodies (ADA)
Description: Serum samples were collected for the determination of anti-GSK3511294 antibodies (ADA) using a validated electro-chemiluminescent immunoassay. The assay involved screening, confirmation and titration assays. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for specificity using the confirmation assay. Samples that confirmed positive in the confirmation assay were reported as 'positive'. Confirmed positive ADA samples were further characterized in the titration assay to quasi-quantitate the amount of ADA in the sample and were also further characterized in the Neutralizing antibody (Nab) assay. A participant was considered positive ADA if they had at least one positive worst case post-Baseline ADA result. Number of participants with worst case post-Baseline positive anti-GSK3511294 antibodies are presented.
Time Frame: Up to Week 52
Population: Safety Analysis Set included all participants who received at least one dose of open-label GSK3511294 excluding the participants from the sites with data integrity and GCP violation issues. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study | GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study
Number analyzed (Participants) | 206 | 416
Participants | 15 | 40

3. Primary Outcome: Number of Participants With Worst Case Post-Baseline Positive Neutralizing Antibodies
Description: Blood samples were collected for the determination of positive neutralizing antibodies. Neutralizing antibody (NAb) test was only carried out on samples that were positive in the confirmatory binding antibody assay. A participant was considered positive for NAb if they had at least one positive worst case post-Baseline neutralizing antibody result. Number of participants with worst case post-Baseline positive neutralizing antibodies are presented.
Time Frame: Up to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study | GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study
Number analyzed (Participants) | 15 | 40
Participants | 0 | 5

4. Secondary Outcome: Annualized Rate of Clinically Significant Exacerbations
Description: Clinically significant exacerbations recorded were defined as worsening of asthma requiring the use of systemic corticosteroids (CS) (such as intramuscular [IM], intravenous [IV] or oral) and/or hospitalization and/or Emergency Department (ED) visit. For all participants, IV or oral steroids (e.g., prednisone) for at least 3 days or a single IM corticosteroid dose is required. For participants on maintenance systemic corticosteroids, at least double the existing maintenance dose for at least 3 days is required. Exacerbations recorded in the electronic case report form (eCRF) were considered as verified clinically significant exacerbations and included in the analysis. Exacerbations separated by less than 7 days was treated as a continuation of the same exacerbation.
Time Frame: Up to Week 52
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Exacerbation per participant per year
Arm/Group | Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study | GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study
Number analyzed (Participants) | 210 | 419
Exacerbation per participant per year | 0.58 [0.45 to 0.73] | 0.55 [0.47 to 0.66]

5. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-5 (ACQ-5) Score
Description: The ACQ-5 is a five-item questionnaire developed as a measure of participants asthma symptom control. The questions are designed to be self-completed by the participant. The 5 questions enquired to recall how their asthma had been during the previous week and to respond about the frequency and/or severity of symptoms (nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheezing). The overall ACQ-5 response option is the mean score of all 5 questions representing 0 with no impairment/limitation and 6 as total impairment/ limitation. Higher scores indicated more limitations and lower score with better asthma control. Baseline was the value at Day 1 of the study. Change from Baseline was defined as value at the indicated time point minus Baseline value. Number of participants with analyzable data for one or more timepoints.
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 20, 26, 28, 32, 40 and 52
Population: Safety Analysis Set included all participants who received at least one dose of open-label GSK3511294 excluding the participants from the sites with data integrity and GCP violation issues. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study | GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study
Number analyzed (Participants) | 195 | 403
Scores on a Scale
  Week 4: number analyzed (Participants) | 179 | 363
  Week 4 | -0.28 (0.056) | -0.16 (0.039)
  Week 8: number analyzed (Participants) | 183 | 384
  Week 8 | -0.22 (0.056) | -0.19 (0.039)
  Week 12: number analyzed (Participants) | 184 | 386
  Week 12 | -0.28 (0.055) | -0.22 (0.038)
  Week 20: number analyzed (Participants) | 183 | 386
  Week 20 | -0.16 (0.058) | -0.16 (0.040)
  Week 26: number analyzed (Participants) | 186 | 393
  Week 26 | -0.14 (0.055) | -0.12 (0.038)
  Week 28: number analyzed (Participants) | 181 | 392
  Week 28 | -0.23 (0.057) | -0.24 (0.039)
  Week 32: number analyzed (Participants) | 187 | 388
  Week 32 | -0.35 (0.057) | -0.25 (0.040)
  Week 40: number analyzed (Participants) | 183 | 383
  Week 40 | -0.24 (0.065) | -0.16 (0.045)
  Week 52: number analyzed (Participants) | 180 | 381
  Week 52 | -0.15 (0.059) | -0.11 (0.041)

6. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score at Weeks 26 and 52
Description: The SGRQ is a 50-item patient-reported outcome tool used to measure Quality of Life in participants with airway obstruction diseases. The questions are designed to be self-completed by the participant. The total score was calculated by the symptom score, activity and impact score; and summarizing the impact of the disease on overall health status on 0-100 rating scale. Scores are expressed as a percentage of overall impairment where 100 representing worst possible health status and 0 indicating best possible health status. Higher scores indicating greater impairment of quality of life. Baseline was the value at Day 1 of the study. Change from Baseline was defined as value at the indicated time point minus Baseline value. Number of participants with analyzable data for one or more timepoints.
Time Frame: Baseline (Day 1), Weeks 26 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study | GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study
Number analyzed (Participants) | 188 | 396
Scores on a Scale
  Week 26: number analyzed (Participants) | 176 | 379
  Week 26 | -5.00 (0.939) | -2.62 (0.641)
  Week 52: number analyzed (Participants) | 174 | 373
  Week 52 | -4.75 (1.043) | -2.33 (0.713)

7. Secondary Outcome: Change From Baseline in Pre-Bronchodilator Forced Expiratory Volume in One Second (FEV1) at Weeks 26 and 52
Description: Forced Expiratory Volume in One Second (FEV1) is a measure of lung function and defined as the volume of air that can be forced out in one second after taking a deep breath. FEV1 was measured electronically by spirometry. Baseline was the value at Day 1 of the study. Change from Baseline in pre-bronchodilator FEV1 was defined as value at the indicated time point minus Baseline value. Number of participants with analyzable data for one or more timepoints.
Time Frame: Baseline (Day 1), Weeks 26 and 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study | GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study
Number analyzed (Participants) | 195 | 402
Liters (L)
  Week 26: number analyzed (Participants) | 193 | 398
  Week 26 | 0.059 (0.0207) | 0.013 (0.0144)
  Week 52: number analyzed (Participants) | 188 | 379
  Week 52 | 0.036 (0.0217) | -0.004 (0.0152)

ADVERSE EVENTS:
Time Frame: Up to Week 56
Description: All-cause mortality, serious adverse events and common non-serious adverse events were reported for the Safety Analysis Set which included all participants who received at least one dose of open-label GSK3511294 in this extension study, excluding the participants from the sites with data integrity and GCP violation issues.
Arm/Group | Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study | GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study
All-Cause Mortality (participants affected / at risk) | 0/210 | 0/419
Serious Adverse Events (participants affected / at risk) | 21/210 | 38/419
Other Adverse Events (participants affected / at risk) | 82/210 | 178/419
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study (N=210) | GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study (N=419)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Adams-Stokes syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Medical device site haematoma (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Chronic rhinosinusitis with nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Hip deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo in Previous Studies/GSK3511294 100 mg SC in Extension Study (N=210) | GSK3511294 in Previous Studies/GSK3511294 100 mg SC in Extension Study (N=419)
Bronchitis (Infections and infestations) | 7 (7) | 22 (23)
COVID-19 (Infections and infestations) | 15 (15) | 28 (29)
Influenza (Infections and infestations) | 7 (7) | 9 (10)
Lower respiratory tract infection (Infections and infestations) | 6 (8) | 13 (16)
Nasopharyngitis (Infections and infestations) | 21 (27) | 58 (73)
Pharyngitis (Infections and infestations) | 8 (10) | 15 (17)
Respiratory tract infection (Infections and infestations) | 3 (4) | 16 (21)
Rhinitis (Infections and infestations) | 8 (11) | 13 (16)
Upper respiratory tract infection (Infections and infestations) | 25 (33) | 45 (60)
Headache (Nervous system disorders) | 7 (8) | 18 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT05243680/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT05243680/SAP_001.pdf